CLINICAL TRIAL: NCT03616951
Title: Response Evaluation Criteria in Metastatic Renal Cell Carcinoma: Improved Assessment of Response and Progression by Spectral-CT
Brief Title: Improved Assessment of Response in Metastatic Renal Cell Carcinoma Using Spectral-CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Frede Donskov, Consultant, Associate Professor, University of Aarhus
Other Study IDs: 151115
Record Dates: First submitted 2018-05-07; First posted 2018-08-06 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Renal Neoplasm With Metastasis; Response Evaluation Criteria in Solid Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of renal cancer in Denmark is approximately 900 new cases per year. Untreated, the 5-year survival rate for metastatic renal cancer (mRCC) is 2%. Development of angiogenesis inhibitors (AI) and check-point immunotherapy (CPI) has improved survival.

Treatment efficacy is evaluated by CT scans, using RESIST 1.1 (Response Evaluation Criteria in Solid Tumors). However, progressin in patients with mRCC treated with AI or CPI is difficult to characterize at the right time, using the RECIST 1.1. Therefore approximately 50 % of the patients are 'lost' to further treatment at the time of progression and die.

The investigators aim to evaluate if functional imaging parameters using spectral CT-techniques can detect treatment failure earlier, or more accurate, than routine CT. This could help us develop a new set of response evaluation criteria for functional imaging, giving a more precise assessment of treatment effect in patients with mRCC treated with AI and CPI.

DETAILED DESCRIPTION:
Response evaluation criteria in metastatic renal cell carcinoma: Improved assessment of response and progression by Spectral CT?

Clinical Background

Renal cancer accounts for 2-3% of all cancers. The incidence of renal cancer in Denmark is approximately 900 new cases per year. Renal cell carcinoma (RCC) arises from the renal parenchyma and is by far the most common type. In 20-30% of all new cases, metastases exist at the time of diagnosis. Up to 25-50 % of patients treated with nephrectomy for localized RCC will eventually develop metastases. Untreated, the 5-year survival rate for metastatic RCC (mRCC) is 2%, and the median survival is 3 months. Within the last 10 years, an increased understanding of kidney cancer biology, and the immune system, has resulted in the development and approval of more than 12 new biological drugs. These are characterized by inhibiting the formation of new blood vessels (angiogenesis inhibitors) or by activating the patient's own immune system to attack the cancer disease (check-point inhibitors). Survival has significantly improved for the patient group with these drugs. The treatment results in control of tumor growth in the majority of patients, for a certain length of time, but should be given continuously, has side effects, and is expensive. In case of disease progression, treatment is changed to another drug. Thus, treatment for mRCC comprises sequential alternating drugs for as long as possible. However, progression is difficult to characterize at the right time and approximately 50 % of the patients are 'lost' to further treatment at the time of progression and die. The investigators therefore need improved diagnostic tools for early or more accurate detection of treatment failure, resulting in appropriate change of therapy at the right time. Routinely, treatment efficacy is evaluated by CT scans at baseline and every 3 months, using the criteria laid out in RECIST 1.1 (Response Evaluation Criteria In Solid Tumors). When interpreting the CT scan, the sizes of target lesions are measured, and an increase in the sum of target lesions by 30%, or the appearance of a new lesion, are interpreted as disease progression. However, the size of the tumor does not necessarily represent biological and physiological changes within the tumor; Tumors treated with angiogenesis inhibitors may show little or no change in tumor size, or may enlarge slowly during therapy, in spite of clinical benefit to the patient and extended time-to-progression. New lesions or tumor enlargement may be seen as part of pseudo-progression in patients treated with check-point inhibitors.

Therefore, the criteria from RECIST 1.1, despite being the best available at the moment, are far from an optimal tool for evaluating response and progression in patients with mRCC treated with biological therapy.

Recent studies from the research group behind the current pH.D. project have shown that functional imaging with Dynamic Contrast Enhanced Computer Tomography (DCE-CT) was able to measure changes in blood flow over time in a single metastasis. Using DCE-CT, the best clinical effect of angiogenesis inhibitor therapy was seen in patients with the greatest decline in blood volume and blood flow, measured after 1 month of treatment compared with baseline. In contrast, patients with low blood volume and low blood flow at baseline had the worst survival, with almost no benefit from treatment, regardless of whether they were treated with angiogenesis inhibitors or immunotherapy.

Based on these results, functional imaging using DCE-CT has the potential to serve as a predictive and prognostic tool in patients with mRCC. However, the DCE-CT technique can only measure functional parameters in one single metastasis and requires use of extra intravenous contrast, and increases radiation dose to the patient.

A new technique, Spectral CT, can visualize and measure functional parameters in all metastases in the body, with use of no extra intravenous contrast, and with no extra radiation dose compared to conventional CT. Spectral CT can quantify parameters such as iodine density and iodine concentration - parameters that could be associated with blood flow and blood volume - and also the relative atomic number can be measured. Response evaluation criteria in metastatic renal cell carcinoma: Improved assessment of response and progression by advanced CT-techniques?

Technical background

Spectral-CT adds spectral resolution to traditional CT scans through a new dual-layer spectral detector. With an Yttrium-based scintillator, the NanoPanel prism detector identifies high-energy and low-energy photons simultaneously, allowing not only anatomy, but also color to characterize the material's content of structures. This new technique allows the characterization of the metastases with parameters such as: iodine density, iodine concentration and the relative atomic number. Spectral CT uses iodinated contrast media -in the same dose as conventional CT. The amount of radiation in a Spectral CT is the same as in a conventional CT.

Aims and hypothesis The present study aims to evaluate functional imaging Spectral-CT as means to improve evaluation of response and progression in patients with mRCC.

The aim is to examine the correlation between Spectral-CT parameters and outcome in patients with mRCC treated with angiogenesis inhibitors and check-point inhibitor immunotherapy.

- Spectral-CT parameters at baseline have predictive and prognostic value, and spectral CT parameters during treatment are more accurate than RECIST 1.1 in determining response and progression.

Materials and Methods The project is an explorative prospective study, in which the investigators will examine the correlation between Spectral-CT functional imaging parameters and outcome in patients with mRCC treated with angiogenesis inhibitors and immunotherapy. CT will be performed at baseline, after 1 and 3 months and then every 3 months until progression or death. CT will be performed using the Spectral IQON scanner from Philips, from which the investigators will receive routine CT images, but also Spectral CT-images. In this way the patients can be their own control. The investigators plan to include 60 patients.

Endpoints and data processing In order to evaluate the accuracy of Spectral-CT imaging, the clinical endpoints best response, progression-free survival (PFS) and overall survival (OS) will be used.

Patient registry

Following patient information will be collected from the patients medical record og registered:

* Demographic data (date of birth, height, weight)
* Information about surgical and non-surgical treatment of renal cell carcinoma
* The patients list of medication
* Localisation of primary tumor and metastasis
* Histological parameters
* Findings on radiological examinations
* Blood tests: hemoglobin, white blood cell count, leucocytes, thrombocytes, creatinin, natrium, potassium, bilirubin, alanine transaminase, alkaline phosphatase, lactate dehydrogenase,calcium, albumine.
* Information about oncologic treatment after the patient progresses in actual study

Ethical Considerations The "Spectral-CT" study is approved by The Central Denmark Region Committees on Health Research Ethics (journal no. 1-10-72-242-17) and is approved the Data Protection Agency (journal no. 1-16-02-791-17). No procedure in the study will be performed before written informed consent has been obtained from each patient.

4. Perspectives Functional imaging using DCE and Spectral CT is considered a potential, new, non-invasive biomarker with the potential to serve as a predictive and prognostic tool. Biomarkers have traditionally been developed by analyzing blood or biopsy material. Core-needle tumor biopsies are, however, invasive procedures with associated discomfort and complications. The development of a non-invasive biomarker, obtained at the same time as routine CT assessment, which has potential for treatment selection (predictive tool) and improved prognostication, would therefore be a significant advance for patient with mRCC. To our knowledge no previous studies have investigated he correlation between DCE-CT parameters and the amount of blood vessels in tumor biopsies. Nor have Spectral CT been used as evaluation of response and progression in mRCC patients. The present study has the potential to develop an updated RECIST - integrating tumor size with functional information. This could give a more precise assessment of oncological treatment, thereby improving patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 18 years
2. Metastatic renal cell carcinoma
3. Oncologic treatment with immunotherapy or angiogenesis inhibitors
4. The patients have signed an informed consent statement
5. Can cooperate for the examinations

Exclusion Criteria:

1. Glomerular filtration fraction below 35 ml/min
2. Allergies or other contraindications to the use of contrast media

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic renal cell carcinoma, who are going to be treated with immunotherapy og angiogenesis inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | PFS is the time from the initiation of therapy and until progressive disease or death, whichever comes first - assessed up to 60 months. If a patient does not progress, PFS will be censored at the time of last follow-up - assessed up to 60 months.
  PFS is the time from the initiation of therapy and until progressive disease or death, whichever comes first, assessed up to 60 months. If a patient does not progress, PFS will be censored at the time of last follow-up - assessed up to 60 months.
overall survival | Overall survival is the time between the first day of treatment and the date of death or last follow-up - assessed up to 60 months.
  Overall survival is the time between the first day of treatment and the date of death or last follow-up - assessed up to 60 months.

SECONDARY OUTCOMES:
Best response | Time from inclusion to best response - assessed up to 60 months.
  Response will be categorized according to the criteria from RECIST 1.1: complete response, partial response, stable disease and progressive disease - assessed up to 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Frede Donskov, MD, DMSc, Principal Investigator — Department of oncology, Aarhus Universety Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drljevic-Nielsen A, Donskov F, Mains JR, Andersen MB, Thorup K, Thygesen J, Rasmussen F. Prognostic Utility of Parameters Derived From Pretreatment Dual-Layer Spectral-Detector CT in Patients With Metastatic Renal Cell Carcinoma. AJR Am J Roentgenol. 2022 May;218(5):867-876. doi: 10.2214/AJR.21.26911. Epub 2021 Dec 15. PMID 34910540